CLINICAL TRIAL: NCT05986656
Title: X-ray Assessment of the Effectiveness of Hardware Medical Acupressure of the Suboccipital Muscles According to the "Atlas-Standard" Method in Patients With Chronic Subluxation of the First Cervical Vertebra
Brief Title: X-ray Evaluation of the Effectiveness of the Atlas Correction in Patients With Chronic Subluxation of the Atlas
Acronym: AtlaStandard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinic of Phlebology and Laser Surgery, Chelyabinsk, Russia (Other)
Responsible Party: Principal Investigator, Denis Borsuk, Director, Clinic of Phlebology and Laser Surgery, Chelyabinsk, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13072023
Record Dates: First submitted 2023-07-16; First posted 2023-08-14 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Subluxation and Dislocation of C0/C1 Cervical Vertebrae
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atlas correction (Experimental): Basic group.
  Interventions: Procedure: Atlas-Standard method

INTERVENTIONS:
Procedure: Atlas-Standard method — Hardware acupressure of the suboccipital muscles according to the Atlas-Standard method for the reduction of chronic subluxation of the first cervical vertebra.

SUMMARY:
The aim of the study is to evaluate the effect of the procedure of medical acupressure of the suboccipital muscles according to the Atlas-Standard method on the normalization of the position of the first cervical vertebra and the angles of the spinal column in patients with diagnosed chronic subluxation with objectification of the results by radiography and inclinometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic subluxation of the first cervical vertebra with complaints of pain in the occiput/cervical/thoracic/lumbar spine/limitation of head rotation in one or both directions.
* Scoliotic deformity of the spine 1-2 degrees.

Exclusion Criteria:

* Pregnancy
* Fractures of the first / second cervical vertebra in history
* Fractures of the spine in any of the departments in the anmenesis
* Assimilation of the atlas with the occipital bone or the second cervical vertebra
* Operations on the spine using metal structures
* Scoliosis 3-4 degree
* Botulinum toxin injections in the suboccipital region within the last year
* Taking muscle relaxants
* Corrective surgery on muscles and bones
* Braces
* Active period of dental implants installation
* Postoperative period (any operation, including on the eyes) less than 6 months
* Acute infectious diseases - less than 2 weeks from the start of recovery
* Skin diseases with inflammatory manifestations in the neck
* Oncological diseases
* Recovery period after injury (cervical and brain injury) or stroke less than a year
* Established mental illness
* Extreme malnutrition (cachexia)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Distance between righr and left inner surface of the lateral mass of the atlas and the outer surface of the odontoid process of the axis on x-ray | 1 month.
  Elimination of asymmetry between the right and left atlantodental intervals

SECONDARY OUTCOMES:
Pain level | 6 month
  Change in the pain level in the spine according to VAS (Visual Analog Scale from 0 to 10 where 0 is "no pain", 10 is "worst pain imaginable")
Painkillers | 6 month
  Number of participants who use painkillers before and after procedure
The functional disability | 6 month
  Evaluated with the Oswestry Disability Index (ODI: 0 = minimal [better outcome] to 100% = maximal disability [worse outcome])
Changes in the angles of deviation of the spinous processes | 6 month
  Measurement of the angles of deviation of the spinous processes in degrees of the frontal and sagittal cavities from C7 to S3 in the position of full flexion, extension of the spine and in the vertical position measured by Spinal Mouse device
Changes in the range of motion of the spine | 6 month
  Changes in the range of motion of the spine in degrees in the frontal and sagittal planes in the range from C7 to S3 in the position of full flexion and extension of the spine measured by Spinal Mouse device

CONTACTS AND LOCATIONS:
Overall Officials: Denis Borsuk, Study Chair — South Ural Medical University
Locations (1):
- Astrakhan Regional Clinical Hospital, Astrakhan, Russia

IPD SHARING:
Plan to Share IPD: No